CLINICAL TRIAL: NCT07231276
Title: Prospective Cohort Study on Pegylated Interferon Alfa-2b in Improving Clinical Cure Rate of Adolescent and Pediatric Patients With Chronic Hepatitis B Virus Infection
Brief Title: Prospective Cohort Study on PEG-IFN-α-2b in Improving Clinical Cure Rate of Pediatric Patients With Chronic Hepatitis B
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-346
Record Dates: First submitted 2025-09-18; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HBV; Chronic Hepatitis B Virus
Keywords: HBV; chronic hepatitis B virus
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Pegylated Interferon Alfa-2b) (Experimental): Subjects in the treatment group will receive pegylated interferon alfa-2b treatment. The dosage will be determined based on height and weight, calculated as 180 μg × body surface area / 1.73 m². The administration method is subcutaneous injection once per week for 48 consecutive weeks. Follow-up visits will be conducted during the treatment period (at Week 4, Week 8, Week 12, Week 24, Week 36, and Week 48) and after the end of treatment (at Week 12 post-treatment and Week 24 post-treatment). The total number of injections administered will not exceed 96.
  Interventions: Drug: Peginterferon alfa-2b Injection
- Observation Group (No Intervention): Subjects in the observation group will receive no drug treatment or be treated with nucleos(t)ide analogs, and will undergo regular follow-up at the specified time points (Week 12, Week 24, Week 48, Week 60, and Week 72).

INTERVENTIONS:
Drug: Peginterferon alfa-2b Injection — Subjects in the treatment group will receive pegylated interferon alfa-2b treatment. The dosage will be determined based on height and weight, calculated as 180 μg × body surface area / 1.73 m². The administration method is subcutaneous injection once per week for 48 consecutive weeks. Follow-up visits will be conducted during the treatment period (at Week 4, Week 8, Week 12, Week 24, Week 36, and Week 48) and after the end of treatment (at Week 12 post-treatment and Week 24 post-treatment). The total number of injections administered will not exceed 96.
  Arms: Treatment Group (Pegylated Interferon Alfa-2b)

SUMMARY:
In this study, comparisons will be made between the treatment group (which will receive pegylated interferon alfa-2b treatment) and the observation group (which will receive no drug treatment or be treated with nucleos(t)ide analogs). The primary objectives are to address the following questions: compare the efficacy evaluation indicators (with clinical cure rate as the primary one) between the pegylated interferon alfa-2b treatment group and the observation group; assess whether pegylated interferon alfa-2b treatment improves the clinical cure rate in patients with chronic hepatitis B virus (HBV) infection aged 3 years and above but under 18 years (adolescents and children); and explore optimized antiviral treatment regimens for adolescents and children with chronic HBV infection. The secondary objectives are to address the following questions: compare the immune response characteristics between adolescents and children with chronic HBV infection who achieved functional cure after pegylated interferon alfa-2b treatment and those who did not; investigate the immune mechanism underlying the achievement of functional cure in adolescents and children with chronic HBV infection treated with pegylated interferon alfa-2b; and identify plasma markers associated with treatment efficacy for predicting therapeutic outcomes.

DETAILED DESCRIPTION:
This study is a prospective, multicenter study. A total of 113 subjects (adolescent and pediatric patients with chronic hepatitis B virus [HBV] infection) were recruited and divided into a treatment group and an observation group. After collecting baseline data from both groups, the treatment group was administered pegylated interferon alfa-2b, while the observation group received no drug treatment or was treated with nucleos(t)ide analogs. Blood samples were collected at different follow-up time points to detect relevant indicators. By comparing the baseline data with follow-up data during treatment, indicators such as HBV DNA negativity rate, HBeAg seroconversion rate, and HBsAg clearance rate were observed in adolescent and pediatric patients with chronic HBV infection. This was done to evaluate whether pegylated interferon alfa-2b treatment improves the clinical cure rate in this patient population and to explore optimized antiviral treatment regimens for adolescent and pediatric patients with chronic HBV infection. Additionally, the immune response characteristics were compared between adolescent and pediatric patients with chronic HBV infection who achieved functional cure after pegylated interferon alfa-2b treatment and those who did not. This comparison aimed to investigate the immune mechanism underlying functional cure achieved by pegylated interferon alfa-2b in adolescent and pediatric patients with chronic HBV infection, as well as to identify plasma markers associated with treatment efficacy for predicting therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years and above but under 18 years;
* Positive for hepatitis B virus (HBV) DNA;
* Positive for hepatitis B surface antigen (HBsAg) (above the lower limit of baseline detection or > 0.05 IU/ml);
* The subject and their guardian(s) understand the study and voluntarily sign the informed consent form (if the guardians are the subject's parents, both parents must sign jointly).

Exclusion Criteria:

* Co-infection with hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV), hepatitis E virus (HEV), or human immunodeficiency virus (HIV);
* Having contraindications to pegylated interferon alfa-2b:

  1. Decompensated hepatitis B cirrhosis;
  2. Subjects with autoimmune liver disease, metabolic liver disease, alcoholic liver disease, malignant tumor, decompensated liver disease, or a history of organ transplantation;
  3. Subjects with severe neurological or psychiatric diseases;
  4. Subjects with severe thyroid dysfunction, antinuclear antibody hyperactivity, or other autoimmune diseases;
  5. Subjects with diabetes mellitus with poor blood glucose control;
  6. Subjects with retinal or fundus lesions;
  7. Subjects with severe heart disease, coronary heart disease, or cerebrovascular disease;
  8. Subjects with poorly controlled epilepsy;
* Adolescent and pediatric subjects with severe renal dysfunction (e.g., creatinine > 1.5 × upper limit of normal [ULN]);
* Subjects deemed unsuitable for enrollment by the investigator(s).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08-08 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of patients treated with PEG-IFN-α-2b (Pegylated Interferon-α-2b) is evaluated based on HBV serological markers and HBV DNA at baseline, during follow-up, and at the follow-up endpoint. | From enrollment to week 24 post-treatment
  Subjects in the treatment group will receive PEG-IFN-α-2b (Pegylated Interferon-α-2b) treatment for a consecutive 48 weeks. Follow-up visits will be conducted during the treatment period (Weeks 4, 8, 12, 24, 36, and 48) and after treatment completion (Weeks 12 and 24 post-discontinuation), with the total number of injections not exceeding 96.
  The efficacy of the treatment for subjects will be mainly evaluated based on the detection results of HBV serological markers (HBsAg、HBsAb、HBeAg、HBeAb、HBcAb) and HBV DNA at time points including baseline, during follow-up, and at the follow-up endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Yongyin Li, doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No